CLINICAL TRIAL: NCT02095899
Title: Effect of Rufinamide on Chronic Postthoracotomy Pain Syndrome. A Prospective, Randomized, Double-blind, Placebo Controlled, Monocenter Study.
Brief Title: Effect of Rufinamide on Chronic Postthoracotomy Pain Syndrome
Acronym: RUFPTPS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor study patient recruitment
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-253
Record Dates: First submitted 2014-02-14; First posted 2014-03-26 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Peripheral Nerve Injuries; Pain
Keywords: Thoracic Surgical Procedures
MeSH Terms: conditions — Peripheral Nerve Injuries; Pain | interventions — rufinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rufinamide (Experimental): - oral Rufinamide administration as ad-on to Oxycodone
  Interventions: Drug: Rufinamide
- Manitol (Placebo Comparator): - oral Placebo administration - as ad-on to Oxycodone
  Interventions: Drug: Rufinamide

INTERVENTIONS:
Drug: Rufinamide — 2x200mg up to max 2x800mg a day Titration over 20days
  Other Names: Inovelon

SUMMARY:
The purpose of this study is to test if rufinamide has an effect on chronic neuropathic pain in patients with a post thoracotomy pain syndrome.

DETAILED DESCRIPTION:
Patients with chronic neuropathic pain after thoracic surgery will be evaluated and treated with oxycodone. Patients with a stable analgesic regimen, not reaching a good pain relief will be randomized to receive Rufinamide (Inovelon)vs. Placebo as an ad-on treatment to oxycodone. Neurophysiological and clinical data will be monitored.

ELIGIBILITY:
Inclusion criteria, Run-In Phase:

* Age: 18-75 years
* Weight: 50 - 100kg
* Height: 155 - 195cm
* Sufficient command of German language
* Patient after thoracotomy
* Pain duration of more than 6 month.
* Diagnosis of Neuropathic Pain (DN4 questionnaire)
* Average baseline mean last week pain intensity =5 on NRS (numerical rating scale)
* Signed and dated informed consent

Inclusion criteria, Treatment Phase:

* Stable analgesic regimen for at least 7 days prior to randomisation
* Patients not reaching a NRS = 3 (numeric rating scale) with the baseline individually dose adjusted treatment (oxycodone).

Exclusion criteria:

* Contraindications to the class of drugs under study, e.g. (rufinamide, oxycodone) known hypersensitivity or allergy this class of drugs
* Hypersensitivity to triazole derivates - antifungal drugs including: fluconazole (e.g. Diflucan®), posaconazole (Noxafil®), itraconazole (Sporanox®), voriconazole (Vfend®)
* Lactose intolerance, galactosemia or galactokinase deficiency, glucose-galactose malabsorption
* Use of topical analgesics, or nerve block of the affected or adjacent dermatomes (less than to 2 weeks prior to the therapy onset visit or during the study period)
* Women who are pregnant or breast feeding; intention to become pregnant during the course of the study, lack of safe contraception, defined as: female subjects of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not willing or able to use any other second (additional) considered sufficiently reliable by the investigator in individual cases. Female subjects who are surgically sterilized/hysterectomized or post-menopausal for longer than 2 years are not considered as being of child bearing potential
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, severe cardiovascular disease, etc)
* Creatinine clearance = 30 ml/min (estimated from serum creatinine using the Cockcroft - Gault formula) were excluded
* Known drug (opiate or other) or alcohol abuse
* Contraindication to the use of oxycodone
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the subject
* Participation in another study with investigational drugs within the 30 days preceding and during the present study
* Enrollment of the investigators, his/her family members, employees and other dependent persons
* Known neurological disease with peripheral manifestations including neuropathy associated with disease such as diabetes
* Known sensory changes from other medical conditions (e.g. infections affecting the investigation areas, post-herpetic neuralgia)
* Epilepsy
* Abnormal electrocardiogram (especially Familial Short QT syndrome)
* Patient having another pain condition with greater pain intensity
* Repeated thoracic surgeries
* Pneumonectomy or chest wall resection
* Bilateral thoracic surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Area of punctuate hyperalgesia immediately after topical capsaicin. | 2h after capsaicin removal
  The primary variable to test is the area of punctuate hyperalgesia after topical capsaicin application in patients treated with rufinamide versus placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Konrad Maurer, MD, Principal Investigator — University Hospital Zurich, Institut of Anaesthesiology
Locations (1):
- University Hospital Zurich, Institut of Anaesthesiology, Zurich, Canton of Zurich, Switzerland